CLINICAL TRIAL: NCT03202875
Title: A Randomized, Double-Blind, Controlled, Single-Dose, 3-Treatment, 3-Period, 6-Sequence Crossover Study to Compare Exposure and Activity of SAR341402 to NovoRapid® and NovoLog® Using the Euglycemic Clamp Technique, in Subjects With Type 1 Diabetes Mellitus
Brief Title: A Study to Compare Pharmacokinetics (PK) and Pharmacodynamics (PD) of SAR341402 to Insulin Aspart in Subjects With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PDY12695; 2012-002355-42 (EudraCT Number); U1111-1127-2950 (Other: UTN)
Record Dates: First submitted 2017-06-27; First posted 2017-06-29 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Test (T) (Experimental): SAR341402: single dose injection
  Interventions: Drug: SAR341402
- Reference 1 (R1) (Active Comparator): NovoRapid®: single dose injection
  Interventions: Drug: Insulin Aspart
- Reference 2 (R2) (Active Comparator): NovoLog®: single dose injection
  Interventions: Drug: Insulin Aspart

INTERVENTIONS:
Drug: SAR341402 — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Arms: Test (T)
Drug: Insulin Aspart — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: NovoRapid®
  Arms: Reference 1 (R1)
Drug: Insulin Aspart — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: NovoLog®
  Arms: Reference 2 (R2)

SUMMARY:
Primary Objective:

To compare exposure and activity of SAR341402 to NovoRapid® and NovoLog®.

Secondary Objective:

To assess the safety and tolerability of SAR341402.

DETAILED DESCRIPTION:
The total study duration for a screened subject will be about 3 - 8 weeks (excluding screening of 2 to 28 days), treatment period of 2 days for each 3 periods (1 overnight stay), a washout period of 5-18 days (preferentially 7 days between consecutive dosing), and an end-of-study visit of 1 day between Days 5 and 14 after the last administration of the investigational product.

ELIGIBILITY:
Inclusion criteria :

* Male or female subjects with diabetes mellitus type 1 for more than one year.
* Total insulin dose of < 1.2 U/kg/day.
* Fasting negative serum C-peptide (< 0.3 nmol/L).
* Glycohemoglobin (HbA1c) ≤ 9%.
* Stable insulin regimen for at least 2 months prior to study.
* Normal findings in medical history and physical examination (cardiovascular system, chest and lungs, thyroid, abdomen, nervous system, skin and mucosae, and musculo-skeletal system), vital signs, electrocardiogram (ECG) and safety lab.

Exclusion criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic (apart from diabetes mellitus type 1), hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness.
* More than one episode of severe hypoglycemia with seizure, coma or requiring assistance of another person during the past 6 months.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month.
* Symptomatic postural hypotension, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥20 mmHg within 3 minutes when changing from supine to standing position.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol.
* Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication, with the exception of insulins, thyroid hormones, lipid-lowering and antihypertensive drugs and if female with the exception of hormonal contraception or menopausal hormone replacement therapy; any vaccination within the last 28 days.
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11-14 (Actual); Primary Completion 2012-12-28 (Actual); Study Completion 2012-12-28 (Actual)

PRIMARY OUTCOMES:
Assessment of PK parameters: maximum plasma concentration (Cmax) | 12 hours
  Maximum plasma concentration (Cmax) of SAR341402, NovoRapid and NovoLog within 12 hours
Assessment of PK parameters: Area under the concentration versus time curve (AUC) | 12 hours
  INS-AUC of SAR341402, NovoRapid, and NovoLog from 0 to 12 hours
Assessment of PK parameter: AUC from dosing to last concentration (AUClast) | 12 hours
  INS-AUClast is AUC from the time of dosing to the last measurable concentration of SAR341402, NovoRapid, and NovoLog from 0 to 12 hours
Assessment of PD parameters: Area under the body weight standardized glucose infusion rate (GIR) | 12 hours
  Area under the body weight standardized glucose infusion rate (GIR) versus time curve from 0 to 12 hours post administration (GIR-AUC0-12)

SECONDARY OUTCOMES:
Assessment of PK: Fractional area under the concentration versus time curve | 12 hours
  INS-AUC0-2 and INS-AUC4-tlast
Assessment of PK: Time to 20 % of INS-AUC | 12 hours
  Time to 20% of AUC (t20%-INS-AUC) within 12 hours
Assessment of PK: time to reach INS-Cmax (INS-tmax) | 12 hours
  INS-tmax within 12 hours
Assessment of PK: time to reach INS-t1/2z (INS-t1/2z) | 12 hours
  INS-t1/2z within 12 hours
Assessment of PD: Fractional area under the body weight standardized GIR versus time curve | 12 hours
  GIR-AUC0-2 and GIR-AUC4-12
Assessment of PD: Time to 20 % of total GIR-AUC0-12h | 12 hours
  Time to 20% of total GIR-AUC0-12h (t20%-GIR-AUC0-12h) within 12 hours
Assessment of PD: Maximum smoothed body weight standardized GIR (GIRmax) | 12 hours
  Maximum smoothed body weight standardized GIR (GIRmax) within 12 hours
Assessment of PD: Time to GIRmax (GIR-tmax) | 12 hours
  Time to GIRmax (GIR-tmax) within 12 hours
Number of adverse events (AEs) | 8 weeks
  Number of patients with treatment emergent AEs and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site 276001, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Kapitza C, Nosek L, Schmider W, Teichert L, Nowotny I. Single-Dose Euglycemic Clamp Study Demonstrating Pharmacokinetic and Pharmacodynamic Similarity Between SAR341402 Insulin Aspart and US- and EU-Approved Versions of Insulin Aspart in Subjects with Type 1 Diabetes. Diabetes Technol Ther. 2020 Apr;22(4):278-284. doi: 10.1089/dia.2019.0351. Epub 2019 Dec 30. PMID 31825248